CLINICAL TRIAL: NCT03199235
Title: Cooking With Iron Ingots: Assessing Feasibility and Natural History of Iron-deficiency Anemia Among Preschool-aged Children in Resource-limited Settings
Brief Title: Iron Fish in Dominican Republic (DR) Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Lucky Iron Fish (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-012631
Record Dates: First submitted 2017-06-07; First posted 2017-06-26 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Iron Deficiency Anemia; Anemia; Iron-deficiency
Keywords: iron intake; iron bioavailability
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIF + Citrus (Experimental): Parents of subjects > 1 year and < 5 years with anemia (Hemoglobin < 11.0 g/dL) are provided the lucky iron fish and citrus along with instructions for use. Followed at regular intervals.
  Interventions: Device: Lucky Iron Fish
- enhanced standard of care (Active Comparator): Parents of subjects > 1 year and < 5 years with anemia (Hemoglobin < 11.0 g/dL) are provided the oral iron supplementation consistent with standard of care, and then followed at regular intervals in addition to any care determined to be necessary by regular provider.
  Interventions: Other: enhanced standard of care

INTERVENTIONS:
Device: Lucky Iron Fish — 200g iron ingot that is placed in boiling water for 10+ minutes, and then removed. The water is then used to eating and drinking.
  Arms: LIF + Citrus
Other: enhanced standard of care — parents of subjects are provided oral iron supplementation per usual clinical care at clinic and followed for their anemia in addition to study visits
  Arms: enhanced standard of care

SUMMARY:
The objective of the study is to assess the acceptability, feasibility, and barriers to Lucky Iron Fish™ (LIF) utilization among families with young children in a Latin American community with a high prevalence of iron deficiency and iron-deficiency anemia.

.

DETAILED DESCRIPTION:
The primary objective is to assess the acceptability of cooking with an iron ingot (Lucky Iron Fish™) compared to traditional oral iron supplementation methods among preschool aged children in a Dominican community with a high prevalence of anemia (> 50%). Data will be collected to characterize the natural history of iron deficiency and anemia in pre-school aged children in a Dominican community. The study will involve a randomized control trial to assess the primary objective: children > 1 year and < 5 years of age will be randomized into two study arms: LIF plus citrus (LIF arm) versus standard iron-supplementation (enhanced standard of care). Participants enrolled in the both study arms will have study labs drawn every 3, 6, and 12-months (hemoglobin, serum ferritin, c-reactive protein) to assess the natural history of iron deficiency in these children. Concomitant to study labs, parents/guardians will be surveyed on acceptability, compliance, and barriers to use of their assigned iron supplementation method.

Primary study outcomes are the change in hemoglobin within the LIF group and then difference in change in hemoglobin between study arms over a 12-month study period. Secondary outcomes include changes in serum ferritin within and between study arms and exploring the relationship between changes in hemoglobin, serum ferritin, and C-reactive protein

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian ≥ 18 years of age
* Child > 1 year and < 5 years of age
* Child followed by Niños Primeros en Salud (NPS)
* Parent/guardian is Spanish speaking
* Parental/guardian permission is provided (informed consent)

Exclusion Criteria:

* Mother/Infant pairs enrolled in related protocol of this study
* Inability to understand and speak Spanish
* Severe cognitive impairment or severe psychiatric disease which would prohibit the answering of study questions
* Child followed by NPS malnutrition program
* Persons receiving pre-designed nutrient-fortified foods or participation in another nutrition program
* Child has documented sickle cell disease

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Rates of refusal | 12-months
  Rates of refusal to participate in study measured as proportion of subjects refusing to enter study compared to total number approached.
Retention | 12-months
  Within each study arm (Iron ingot vs. Oral iron supplementation), will calculate proportion lost to follow-up. Number of subjects lost to follow up divided total number of subjects enrolled at study entry.
Adherence to iron ingot use | 12-months
  Using a questionnaire with several likert-scale questions, we will assess adherence to iron ingot use. Questions include "When was the last time you used the Fish", "how often do you use the fish for meal preparation", "how often do you use the fish to prepare water", "how long do you typically boil the fish". The answer to each question has between 4-5 possible ordinal responses which will be converted into numerical data (1,2,3,4,5) and cumulative scores will be created to assess degree of use/adherence.
Adherence to oral iron use | 12-months
  Using a questionnaire with several likert-scale questions, we will assess adherence to oral iron supplementation. Questions include: "How many doses were missed each week", "Do you recall dose and frequency of oral iron you were prescribed", "If doses were missed, was this accidental, intentional, or both". The answer to each question has between 4-5 possible ordinal responses which will be converted into numerical data (1,2,3,4,5) and cumulative scores will be created to assess degree of use/adherence.
Natural history of hemoglobin among those subjects using iron ingot | Will be at 4 individual points over a 12-mo period - at enrollment, 3-month follow-up, 6-month follow-up, and 12-month follow-up which is study end. Thus, the time frame is 4 separate visits over a 12-month period
  We will assess changes in hemoglobin WITHIN iron ingot study arm. Hemoglobin will be measured in grams per deciliter (g/dL) and measured at enrollment, 3-months, 6-months, and 12-months. If data is normally distributed, a paired/dependent t-test will be used, if non-normal, a non-parametric test like Wilcoxon's Matched pairs test will be used.
Natural history of hemoglobin among those subjects using oral iron | Will be at 4 individual points over a 12-mo period - at enrollment, 3-month follow-up, 6-month follow-up, and 12-month follow-up which is study end. Thus, the time frame is 4 separate visits over a 12-month period
  We will assess changes in hemoglobin WITHIN oral iron study arm. Hemoglobin will be measured in grams per deciliter (g/dL) and measured at enrollment, 3-months, 6-months, and 12-months. If data is normally distributed, a paired/dependent t-test will be used, if non-normal, a non-parametric test like Wilcoxon's Matched pairs test will be used.
Natural history hemoglobin: Iron ingot vs. Oral iron | 12-month.
  The difference in change in hemoglobin (measure in g/dL) between the study study arms (iron ingot arm vs. oral iron supplementation arm) will be assessed using two-sample t-test (normal distribution) or Wilcoxon-rank-sum (non-normal distribution).

SECONDARY OUTCOMES:
Natural history of serum ferritin among subjects using iron ingot | Will be at 4 individual points over a 12-mo period - at enrollment, 3-month follow-up, 6-month follow-up, and 12-month follow-up which is study end. Thus, the time frame is 4 separate visits over a 12-month period
  We will assess changes in serum ferritin WITHIN iron ingot study arm. Serum ferritin will be measured in nanograms per milliliter (ng/mL) and measured at enrollment, 3-months, 6-months, and 12-months. If data is normally distributed, a paired/dependent t-test will be used, if non-normal, a non-parametric test like Wilcoxon's Matched pairs test will be used.
Natural history of serum ferritin among subjects using oral iron | Will be at 4 individual points over a 12-mo period - at enrollment, 3-month follow-up, 6-month follow-up, and 12-month follow-up which is study end. Thus, the time frame is 4 separate visits over a 12-month period
  We will assess changes in serum ferritin WITHIN oral iron supplementation study arm. Serum ferritin will be measured in nanograms per milliliter (ng/mL) and measured at enrollment, 3-months, 6-months, and 12-months. If data is normally distributed, a paired/dependent t-test will be used, if non-normal, a non-parametric test like Wilcoxon's Matched pairs test will be used.
Natural history serum ferritin: Iron ingot vs. Oral iron | 12-months
  The difference in change in serum ferritin (measured in ng/mL) between the study study arms (iron ingot arm vs. oral iron supplementation arm) will be assessed using two-sample t-test (normal distribution) or Wilcoxon-rank-sum (non-normal distribution).

CONTACTS AND LOCATIONS:
Locations (1):
- Ninos Primeros en Salud, Consuelo, San Pedro de Macorís, Dominican Republic